CLINICAL TRIAL: NCT06993402
Title: DESI- Düsseldorfer ESD Register Study
Brief Title: DESI - Düsseldorfer ESD Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Torsten Beyna (Other)
Responsible Party: Sponsor-Investigator, Torsten Beyna, Head of the Medical Clinic and Gastroenterology, Evangelisches Krankenhaus Düsseldorf
Organization: Evangelisches Krankenhaus Düsseldorf (Other)
Other Study IDs: DESI
Record Dates: First submitted 2024-12-02; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-12

CONDITIONS: Oesophageal Tumour; Gastric Tumours; Duodenal Tumours; Colon Tumours; Rectal Tumours
Keywords: ESD
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Safety and effectiveness of endoscopic submucosal dissection

DETAILED DESCRIPTION:
Background and study objective The standard of care for premalignant and malignant mucosal lesions in the gastrointestinal track with limited submucosal invasion is an endoscopic resection. A curative resection of the neoplasia often necessitates an en-bloc resection, where the resection ends within healthy tissue (R0 resection). Endoscopic submucosal dissection (ESD) is a highly sophisticated resection technique for lesions in the oesophagus, stomach, duodenum, colon and rectum. Multiple studies in Asia already established the safety and efficacy of ESD. In several spezialized centres in the western world the ESD already replaced the endoscopic mucosal resectiona (EMR) as standart of care. The en-bloc resection facilitates an exact histopathological evaluation, thus leading to lower recurrence rates. Besides specified mucosal lesions, there is an increase in the use of ESD to resect expansive and submucosal lesions. Specialised centres like Evangelisches Krankenhaus Düsseldorf have a high number of ESD cases and use ubiquitous in the gastrointestinal tract. Besides the many advantages over EMR there is still the risk of peri- and postinterventional complications with ESD due to the highly demanding technique and the longer procedure duration. This is why patient selection is crucial factor (in this study). To evaluate the safety and efficacy of ESD more prospective data analysis in western centres are necessary. This data will be useful to develop new approaches to improve the method concerning safety and efficacy and patient selection.

ELIGIBILITY:
Inclusion Criteria:

* signed consent form
* Indication for an ESD in the oesophagus, stomach, duodenum, colon or rectum
* Age >18 years

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epithelial gastrointestinal lesions who receive an endoscopic submucosal dissection in the oesophagus, stomach, duodenum, colon or rectum in accordance with the guidelines (or according to the individual decision of the interdisciplinary tumour conference).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | during the procedure
  TSR, defined as rate of procedures with endoscopic en-bloc resection
Complication rate | through study completion, an average of 5 years
  Serious complications, (according to AGREE criteria), intraprocedural or late onset
Histopahological result | up to 14 days after Procedure
  Histopathological result of R0 resection (margins are clean, vertical and lateral)

SECONDARY OUTCOMES:
Complete resection rate (endoscopic) | up to 14 days after Procedure till histopathological results
Clinical success rate (curative resection according to standard of care guidelines) | up to 14 days after Procedure till histopathological results
Enhances clinical success rate (no curative resection according to standard of care guidelines, but no further treatment necessary (after individual discussion of cases in tumorboard) | about 4 weeks after the ESD
Complication rate (total) | through study completion, an average of 1 year
Contributing factors on the technical and clinical success rate originating with patient and investigator aspects | through study completion, an average of 1 year
Dissection speed and rate of complications with different ESD devices | during the procedure / 1 day
Recurrence rate after 3, 6, 12, 24 and 60 months (if available) | through study completion, an average of 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Torsten PD Dr. med Beyna, Principal Investigator — Evangelisches Krankenhaus Düsseldorf
Locations (1):
- Evangelisches Krankenhaus Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No